CLINICAL TRIAL: NCT01246518
Title: An Open, Multi-centre Trial Comparing the Efficacy and Safety of Two Different Treatment Regimens of Topical MOB015 Treatment of Distal Subungual Onychomycosis (DSO)
Brief Title: Efficacy and Safety of Two Treatment Regimens of Topical MOB015 in Adults With Distal Subungual Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Kjell Rensfeldt MD, Moberg Derma AB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOB015-I
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2011-09

CONDITIONS: Onychomycosis
Keywords: distal subungual onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOB015 for 3 months (Active Comparator)
  Interventions: Drug: MOB015
- MOB015 for 9 months (Active Comparator)
  Interventions: Drug: MOB015

INTERVENTIONS:
Drug: MOB015 — Arm 1; MOB015 once a day for 3 months. Arm 2; MOB015 once a day for 9 months.

SUMMARY:
Onychomycosis is a fungal infection that affects fingernails and/or toenails.

The purpose of this trial is to investigate if MOB015 is effective and safe for treatment of patients with fungal infection of the toenails.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 18 - 70 years
3. DSO of at least one of the great toe(s) affecting 25 % to 75 % of the target nail (verified by blinded assessor before randomization)
4. Positive culture for dermatophytes (i.e. Trichophyton species; T. rubrum or T. mentagrophytes)
5. Signed written informed consent

Exclusion Criteria:

1. Proximal subungual onychomycosis
2. DSO of both great toenails where involvement has extended into the proximal portion of the target nail (unaffected proximal nail is less than 2 mm)
3. "Spike" of onychomycosis extending to eponychium of the target nail
4. Presence of dermatophytoma (defined as demarcated and localised thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail
5. Other conditions than DSO known to cause abnormal nail appearance
6. Topical antifungal treatment of the nails within 1 month before screening
7. Systemic use of antifungal treatment within 3 months before screening
8. Signs of severe peripheral circulatory insufficiency
9. Immunosuppression
10. Participation in another clinical trial with an investigational drug or device during the previous 4 weeks before screening
11. Known allergy to any of the tested treatment products
12. A pregnancy test indicating pregnancy in a woman of childbearing potential at screening (visit 1)
13. Pre-menopausal (last menstruation ≤ 1 year prior to screening) sexually active women who :

    * are pregnant or nursing
    * are not surgically sterile
    * are of child bearing potential and not practising an acceptable method of birth control, or does not plan to continue practising an acceptable method of birth control throughout the trial (acceptable methods include intrauterine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mycological cure of target nail at 12 months, defined as negative fungal culture and negative direct microscopy. | 12 months

SECONDARY OUTCOMES:
Proportion of patients with negative fungal culture, negative direct microscopy and complete cure. | 1, 3, 6, 9, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Faergemann, MD, PhD, Principal Investigator — Dept. of Dermatology, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- 15 Locations, Sweden, Sweden